CLINICAL TRIAL: NCT02272270
Title: Phase 1 Trial in Newly Diagnosed High Grade Glioma With Temozolomide, Radiation, and Minocycline Followed by Adjuvant Minocycline/Temozolomide. (D-TERMINED)
Brief Title: Phase I Newly Diagnosed GBM With Temozolomide, Radiation, and Minocycline Followed by Adjuvant Minocycline/Temozolomide (D-TERMINED)
Acronym: D-TERMINED
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCI75289
Record Dates: First submitted 2014-10-20; First posted 2014-10-22 (Estimated); Last update posted 2019-06-19 (Actual); Status verified 2019-06

CONDITIONS: Newly Diagnosed High Grade Glioma
MeSH Terms: interventions — Minocycline; Chemoradiotherapy; Temozolomide; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment with Study Agent Combination (Experimental): Radiation Therapy 2.0GyX30fx, 5 days per week for a total of 60 Gy Temozolomide 75mg/m2 daily throughout radiation Minocycline begins one week prior to chemoradiation, and continues twice a day throughout radiation Arm -2:100mg PO BID Arm -1:150mgPO BID Arm 0: 200mg PO BID Arm 1: 400mg PO BID Arm 1a: 300mg PO BID
  Followed by 28 day break followed by
  Temozolomide 150-200mg/m2 on days 1-5 out of 28 for up to12 cycles
  Minocycline taken twice a day throughout each 28 day cycle for up to 12 cycles:
  Arm -2:100mg PO BID Arm -1:150mgPO BID Arm 0: 200mg PO BID Arm 1: 400mg PO BID Arm 1a: 300mg PO BID
  Interventions: Drug: Minocycline with chemoradiation (temozolomide and radiation therapy)

INTERVENTIONS:
Drug: Minocycline with chemoradiation (temozolomide and radiation therapy) — Patients receive minocycline in conjunction with standard chemoradiation and then they receive minocycline with standard chemotherapy.

SUMMARY:
This will be an open label, single arm study. Subjects with newly diagnosed high grade glioma will begin minocycline one week prior to beginning postoperative chemoradiation and continue it until progression, intolerance, or the end of adjuvant temozolomide, whichever comes first.

ELIGIBILITY:
Inclusion Criteria:

Male or female patients greater than or equal to 18 years old Histopathologically proven diagnosis of glioblastoma (GBM) or gliosarcoma or anaplastic astrocytoma(AA) A diagnostic contrast-enhanced MRI or CT scan of the brain must be performed preoperatively and postoperatively (preferably within 96 hours of surgery), prior to the initiation of radiotherapy. The post-operative MRI must be within 35 days prior to study registration.

Patients unable to undergo MR imaging because of non-compatible devices can be enrolled, provided pre- and post-operative contrast-enhanced CT scans are obtained and are of sufficient quality.

Radiation therapy planned to start less than or equal to 6 weeks after surgery and at least 7 days after the start of minocycline Women of child-bearing potential must have a negative pregnancy test within 7 days of initiation of dosing and must agree to use an acceptable method of birth control while on study drug and for 3 months after the last dose. Women of non-childbearing potential may be included if they are either surgically sterile or have been postmenopausal for greater than or equal to1 year. Men of child-bearing potential must also agree to use an acceptable method of birth control while on study drug, and for 3 months after the last dose.

Karnofsky performance status of greater than or equal to 70 Adequate bone marrow function, coagulation, hepatic, and renal function as defined by lab testing.

Exclusion Criteria:

Prior radiation or chemotherapy for high grade glioma Prior invasive cancer (except nonmelanoma skin cancer) unless disease free for at least 2 years or life expectancy without treatment is greater than 2 years, e.g., low risk localized prostate cancer.

Prior radiation to the head or neck with overlapping radiation fields Patients who had a stereotactic needle biopsy Unstable angina and/or decompensated congestive heart failure in the last 6 months, transmural myocardial infarction within the last 6 months, New York Heart Association grade II or higher congestive heart failure requiring hospitalization within 12 months prior to registration, serious or inadequately controlled cardiac arrhythmia, significant vascular and peripheral vascular disease, evidence of bleeding diathesis or coagulopathy.

History of stroke, cerebral vascular accident (CVA) or transient ischemic attack within 6 months Active (acute or chronic) or uncontrolled severe infections requiring intravenous antibiotics Liver disease such as cirrhosis, chronic active hepatitis or chronic persistent hepatitis Acquired immune deficiency syndrome (AIDS) based upon current CDC definition or known HIV seropositivity; note, however, that HIV testing is not required for entry into this protocol. The need to exclude patients with HIV/AIDS from this protocol is necessary because the treatments involved in this protocol may be significantly immunosuppressive.

Active connective tissue disorders, such as lupus or scleroderma Patients with history of allergic reaction to minocycline or to any of the tetracyclines Patients with history of erosive esophagitis should be excluded from the study Patients that are on anticonvulsant medications would be switched, when possible, to a non-enzyme-inducing antiepileptic drug (non-EIAED). However, if that is not possible, they will not be excluded from the study.

Other major medical illnesses or psychiatric impairments that in the investigator's opinion will prevent administration or completion of protocol therapy Women who are breast feeding, due to possible adverse effects on the infant Prior allergic reaction to temozolomide

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2014-10-27 (Actual); Primary Completion 2017-03-08 (Actual); Study Completion 2018-02-18 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of minocycline combined with standard radiation and chemotherapy | Patient safety will be evaluated throughout the treatment period (treatment with Temozolomide, Radiation, and Minocycline followed by Adjuvant Minocycline/Temozolomide) which is expected to last about and up to 14 months for each patient
  The adverse event rate and maximum tolerated dose of minocycline (up to a maximum dose of 800 mg/day) when combined with concurrent radiation and temozolomide in newly diagnosed high grade glioma is being explored.

CONTACTS AND LOCATIONS:
Locations (1):
- Huntsman Cancer Institute, Salt Lake City, Utah, United States